CLINICAL TRIAL: NCT05600686
Title: A Phase 2 Study of Loncastuximab Tesirine and Rituximab (Lonca-R) Followed by DA-EPOCH-R in Previously Untreated High-Risk Diffuse Large B-Cell Lymphoma
Brief Title: Loncastuximab Tesirine and Rituximab Followed by DA-EPOCH-R for Treating Patients With High-Risk Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Joseph Tuscano (Other)
Collaborators: National Cancer Institute (NCI) (NIH); ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor-Investigator, Joseph Tuscano, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#303; NCI-2022-07762 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC#303 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2022-10-10; First posted 2022-10-31 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Double-Expressor Lymphoma; High Grade B-Cell Lymphoma With MYC and BCL2 and/or BCL6 Rearrangements; High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements
MeSH Terms: interventions — Cyclophosphamide; Doxorubicin; Etoposide; loncastuximab tesirine; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Lonca-R, DA-EPOCH-R) (Experimental): Patients receive rituximab IV, loncastuximab tesirine IV, etoposide IV, doxorubicin IV, vincristine IV, prednisone PO, and cyclophosphamide IV on study. Patients also undergo collection of blood samples and bone marrow aspiration and biopsy at screening and CT or PET/CT at screening, throughout the study, and during follow up.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Etoposide; Biological: Loncastuximab Tesirine; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Biological: Loncastuximab Tesirine — Given IV
  Other Names: ADC ADCT-402; ADCT-402; Anti-CD19 PBD-conjugate ADCT-402; Loncastuximab Tesirine-lpyl; Zynlonta
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima
Drug: Vincristine — Given IV
  Other Names: Leurocristine; VCR; Vincrystine

SUMMARY:
This phase II trial evaluates whether loncastuximab tesirine and rituximab followed by dose-adjusted doxorubicin, etoposide, vincristine, cyclophosphamide, and prednisone works to treat patients with high risk diffuse large B-cell lymphoma. Loncastuximab tesirine is a monoclonal antibody called loncastuximab, linked to a drug called tesirine. It is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, known as CD19 receptors, and delivers tesirine to kill them. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Chemotherapy drugs such as doxorubicin, vincristine, and cyclophosphamide work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Etoposide is in a class of medications known as podophyllotoxin derivatives. It blocks a certain enzyme needed for cell division and DNA repair and may kill cancer cells. Prednisone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response to help lessen the side effects of chemotherapy drugs. Giving loncastuximab tesirine and rituximab in combination with dose-adjusted doxorubicin, etoposide, vincristine, cyclophosphamide, and prednisone may be more effective at treating high risk diffuse large B-cell lymphoma patients than standard treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To obtain a preliminary estimate of the anti-tumor activity of loncastuximab tesirine and rituximab (lonca-R) in newly diagnosed double-expressor lymphoma (DEL) and double-hit lymphoma (DHL).

SECONDARY OBJECTIVES:

I. To obtain additional efficacy measures of lonca-R in newly diagnosed DEL and DHL.

II. To assess safety and tolerability of lonca-R followed by dose-adjusted doxorubicin, etoposide, vincristine, cyclophosphamide, and prednisone (DA-EPOCH-R) as coded by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.

OUTLINE:

Patients receive rituximab intravenously (IV), loncastuximab tesirine IV, etoposide IV, doxorubicin IV, vincristine IV, prednisone orally (PO), and cyclophosphamide IV on study. Patients also undergo collection of blood samples and bone marrow aspiration and biopsy at screening and computed tomography (CT) or positron emission tomography (PET)/CT at screening, throughout the study, and during follow up.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed untreated DEL and DHL diffuse large B-cell lymphoma (DLBCL) meeting the World Health Organization (WHO) criteria for DEL - MYC greater than 40% and BCL2 greater than 50% by immunohistochemistry, or high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements (double-hit and/or triple-hit are included)
* Measurable disease by CT or PET/CT scan, with one or more sites of disease >= 1.5 cm in longest dimension
* Age >= 18 years at time of consent
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy >= 6 months
* Leukocytes >= 2,500/uL
* Absolute neutrophil count >= 1,000/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 8 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level =< 3 x ULN may be enrolled)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN (AST and/or ALT =< 5 x ULN for patients with liver involvement)
* Alkaline phosphatase =< 2.5 x ULN (=< 5 x ULN for patients with documented liver involvement or bone metastases)
* Creatinine clearance >= 30 mL/min by Cockcroft-Gault
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN (This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation, such as low-molecular-weight heparin or warfarin, should be on a stable dose)
* Transthoracic echocardiography (TTE) or multigated acquisition scan (MUGA) ejection fraction greater than 40%
* Women of child-bearing potential (WOCBP) must agree to use a highly effective method of contraception from the time of giving informed consent until at least 10 months after the last dose of study drug. Men with female partners who are of childbearing potential must agree to use a highly effective method of contraception from the time of giving informed consent until at least 7 months after the last dose of study drug
* Ability to understand and the willingness to sign a written informed consent document
* Human immunodeficiency virus (HIV) infected patients:

  * No history of acquired immunodeficiency syndrome (AIDS)-defining conditions other than lymphoma or history of CD4+ T-cells below 200/mm^3 prior to beginning combination anti-retroviral therapy (ART)
  * Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
  * At time of study entry CD4+ T-cells must have recovered from prior lymphoma therapy to >= 250/mm^3
  * At the time of study entry, the HIV viral load must be undetectable by standard laboratory assay
  * During prior lymphoma therapy, patients must not have experienced documented infections attributed to the HIV positive (+) status
  * No history of non-adherence to ART and willing to adhere to ART while on study
  * Antiretroviral drugs with overlapping or similar toxicity profiles as study agents not allowed

Exclusion Criteria:

* Current/ prior use of:

  * Lymphoma treatment, except for:

    * 1 cycle of DA-EPOCH-R or rituximab, cyclophosphamide, doxorubicin (Adriamycin) vincristine (Oncovin) and prednisolone (R-CHOP)
    * Radiotherapy > 2 weeks of initiating study treatment
    * Nitrosoureas or mitomycin C > 6 weeks of initiating study treatment
    * Steroid treatment for DLBCL or steroid monotherapy to stabilize disease while awaiting fluorescence in situ hybridization (FISH)
    * Other cancer therapies (e.g., prostate, breast hormonal-based therapy) per the principal investigator's discretion
  * Anthracycline greater than 50 mg/m^2 (total lifetime) for a prior malignancy
  * Complementary and alternative medications (CAM) within 1 week prior to initiating study treatment
  * Treatment with any other investigational agent for any indication within 3 weeks prior to initiating study treatment
  * Loncastuximab tesirine or rituximab with progression within 6 months of initiating study treatment
  * Oral or intravenous (IV) antibiotics within 2 weeks prior to initiating study treatment. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
  * Live, attenuated influenza vaccine within 4 weeks prior to initiating study treatment
* Immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor, such as anti-tumor necrosis factor [TNF] agents) within 14 days prior to initiating study treatment. The following are exceptions to this criterion:

  * Steroids
  * Bisphosphonate therapy for symptomatic hypercalcemia or for other reasons (e.g., bone metastasis or osteoporosis)
* Known uncontrolled central nervous system (CNS) involvement by lymphoma, including leptomeningeal involvement
* History of hypersensitivity to anti-CD19 antibodies, loncastuximab tesirine, or any agents used in DA-EPOCH-R
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to other agents used in study
* Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath)
* Breastfeeding or pregnancy
* Clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; or inherited liver disease

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HbsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* Documented eczema, psoriasis, or lichen simplex chronicus of vitiligo with dermatologic manifestations (e.g., patients with psoriatic arthritis would be excluded), unless the following apply:

  * Affected skin covers less than 10% of body surface area (BSA)
  * Disease is well controlled at baseline and only requires low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
  * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* Known active tuberculosis (TB)
* Severe infections within 4 weeks prior to initiating study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Major surgical procedure within 28 days prior to initiating study treatment or anticipation of need for a major surgical procedure during the course of the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | First dose through cycle 2 (1 cycle = 3 weeks)
  Evaluated per 2014 Lugano criteria. An exact 95% confidence interval will be calculated.

SECONDARY OUTCOMES:
Overall survival rate | First dose to off study, assessed up to 3 years
  Will be estimated using the product-limit of Kaplan and Meier.
Relapse/progression free survival | First dose (cycle 1 day 6 rituximab dose) until relapse/progression or off study, whichever occurs first, assessed up to 3 years
  Will be estimated using the product-limit of Kaplan and Meier.
Overall response rate (complete response + partial response) | First dose through cycle 2 (1 cycle = 3 weeks)
  Defined as the proportion of participants who have partial or complete response from the start of study treatment through completion of 2 cycles. Evaluated per 2014 Lugano criteria. An exact 95% confidence interval will be calculated.
Incidence of adverse events | First dose through 30 days post last dose
  Will evaluate the number of participants experiencing treatment-related adverse events, classified by severity and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Observed toxicities will be summarized by type (organ affected or laboratory determination), severity, date of onset, duration, and attribution.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Tuscano, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Diego Moores Cancer Center, San Diego, California